CLINICAL TRIAL: NCT06547372
Title: Dietary Intervention on Atopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, CHEW Fook Tim, Associate Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUS-IRB-2024-28
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis; Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Throughout the 2-month intervention period, only participants in the intervention arm will be provided with bento-styled meals for lunch and dinner daily. The meals will encompass a variety of nutrient-rich ingredients, including whole grains, lean proteins, an array of fruits and vegetables, and healthy fats. The food will be prepared by a licensed food catering service.
  Interventions: Other: Dietary Intervention on Atopy
- Control (No Intervention): The control group will not receive the meals provided by our study nor will they receive any nutritional advice. Instead, they will continue following their usual dietary habits and patterns throughout the study period.

INTERVENTIONS:
Other: Dietary Intervention on Atopy — The primary aim of this dietary intervention study is to assess the effectiveness of a dietary pattern characterized by lower saturated fats, higher wholegrains, fruit, and vegetables in reducing the severity of AD in young Singapore adults, as measured by changes in Scoring Atopic Dermatitis (SCORAD) scores, over a 2-month intervention period.
  Arms: Intervention

SUMMARY:
Dietary habits play an indispensable role in maintaining overall health and well-being. In recent years, emerging research has underscored the importance of dietary factors on a range of diseases which include allergic (atopic) diseases such as atopic dermatitis (AD). Conducting a dietary intervention study related to AD can provide valuable insights into the relationship between diet and the development or management of this particular allergic skin condition.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic inflammatory skin disease highly associated with xerosis and pruritus, affecting a substantial portion of individuals of all age groups. The European Academy of Allergy and Clinical Immunology (EAACI) Task Force on Diet and Immunomodulation also emphasized the role of dietary patterns as an important indicator to study the risk of allergic diseases. Furthermore, emerging epidemiological findings and randomised controlled trials (RCT) in recent decades strongly suggest that diet may play a pivotal role in not only triggering and exacerbating AD but also in its effective management.

Preliminary cross-sectional findings in a large independent allergic cohort of 13,561 young Chinese Adults from Singapore and Malaysia highlighted that a frequent intake of high-fat foods such as margarine, butter, seafood, and burgers and fast foods is strongly associated with a higher risk of AD. A diet consisting mainly of high-fat foods, or a high-fat diet as shown by a derived amount- and score-based dietary indices was strongly associated with a higher risk for severe AD even controlling for potential confounding factors like age, sex, body mass index (BMI), lifestyle habits, and genetic predisposition. On the other hand, a frequent adherence to a plant-based food dietary pattern consisting of fruit, vegetables, and cereals was associated with a lowered risk of severe AD. Overall, these compelling findings aligned with evidence-based guidelines such as "My Healthy Eating Plate, Singapore", a visual guide designed to promote a balanced and nutritious dietary pattern specific to the Singaporean context.

In conclusion, a whole diet dietary intervention on AD that adhere to established dietary recommendations such as "My Healthy Eating Plate, Singapore", may offer a promising avenue for individuals seeking to i) improve AD symptoms, ii) improve skin health, and iii) improve quality-of-life.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of current, mild-to-moderate atopic dermatitis/eczema at flexural areas
2. 21 to 65 years of age (inclusive) at screening
3. Must be English-literate and able to give informed consent in English
4. Be residing in Singapore and will not be travelling outside of Singapore during the study period
5. Reliable and willing to follow study procedures and be available for the duration of the study
6. Non-smokers (tobacco and e-cigarette)
7. Non-drinker (no regular or frequent consumption of alcohol)
8. Overtly healthy with no pre-existing medical conditions (e.g., diabetes, hypertension, cancer, blood disorders, degenerative/liver/autoimmune/immune/renal diseases, or psychiatric conditions)
9. No food allergies to test foods
10. No needle phobia
11. Be willing to not apply any moisturiser, cosmetics, and/or topical cream on the skin throughout the entire duration of the study.

Exclusion Criteria:

1. Concurrent participation in other research studies
2. Pregnancy or lactating individuals
3. Known or ongoing psychiatric disorders within 3 years
4. Known severe nutritional deficiency
5. Vegetarian/vegans (as meat will be included in the diet)
6. Individuals who made a significant dietary change in the past 12 months
7. Having a pre-existing dietary restriction that would interfere with the adherence to a whole diet meal
8. Regular use of strong medication (western and/or traditional), therapies, and alternative medications
9. Regular nutritional supplements in the past 12 months Regular consumption of oral contraceptive pills and/or steroid hormones
10. Antibiotic use in the past 2 months
11. Any long-term hospitalisation or surgery during the 6 months before enrolment in study
12. Significant change in weight (+/- 5.0%) during the past month
13. History of bleeding diathesis or coagulopathy (or any bleeding disorders)
14. Having donated blood of more than 500 mL within 4 weeks of study enrolment

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of SCORAD Scores by a Healthy Dietary Pattern | 3 months
  To assess the effectiveness of a dietary pattern characterized by lower saturated fats, higher wholegrains, fruit, and vegetables in reducing the severity of AD in young Singapore adults, as measured by changes in Scoring Atopic Dermatitis (SCORAD) scores, over a 2-month intervention period.
  The SCORAD index, a comprehensive and validated tool, is used to assess AD severity by incorporating objective measures of skin lesions, subjective symptoms, and affected body surface extent. SCORAD will assess the percentage of AD in specific body parts (head, neck, limbs, trunk, back) and evaluate the extent and severity of AD by examining erythema, edema, oozing/crusts, excoriation, lichenification, and dryness.SCORAD's standardized and quantitative assessment facilitates accurate baseline characterization and precise monitoring of changes during the intervention.

SECONDARY OUTCOMES:
To determine the impact of an improved dietary pattern on the quality of life of participants with AD, using the Dermatology Life Quality Index (DLQI) in reducing the severity of AD in Singapore adults | 3 months
  The DLQI serves as a valuable metric to gauge the psychological impact of AD on individuals' daily lives. As AD not only affects the skin but also the overall well-being, assessing the intervention's influence on participants' quality of life (QOL) is essential. By incorporating DLQI alongside SCORAD scores, it can comprehensively evaluate the holistic effects of the improved dietary pattern intervention.
  DLQI is computed by assigning scores to 10 questions related to the impact of skin disease on different aspects of daily life, with a total score ranging from 0 to 30, where higher scores indicate a greater impairment of QOL. A DLQI score of 4 is recommended for the threshold for MCID even though it varies from 3 to 5.
Number of participants with improved skin barrier functions as assessed by skin hydration, transpidermal water loss, pH, and sebum level | 3 months
  Measuring skin parameters provides an objective evaluation of the physiological aspect of AD. Each AD participant will be assessed using four bioengineering devices: Tewameter® (measuring transepidermal water loss (TEWL) in g/h/m² by the density gradient of water evaporation), Corneometer® (measuring relative permittivity (F/m) of upper skin layers), Skin-pH-Meter PH® (measuring skin surface pH on a scale of 1-11), and Sebumeter® (measuring sebum content in units from 0-350 based on light transmission through a special tape). Measurements will be taken from predetermined areas assessed using SCORAD.
Number of participants with changes in immune functions as assessed by blood cytokine and chemokine levels. | 3 months
  Participants in the intervention group will follow a specified dietary pattern, while the control group will maintain regular dietary habits. A total of 5mL whole blood samples will be collected and multiplex assays will then be conducted to analyze multiple cytokines simultaneously in each sample.
Number of participants with changes in gene expression profile as assessed by the changes in differentially expressed genes (DEGs). | 3 months
  Examining gene expression changes in response to an improved dietary pattern in AD can reveal potential molecular targets, offering insights into personalized treatment and the link between genetics and diet in AD pathogenesis. Functional enrichment analysis will further elucidate the biological processes, pathways, and molecular functions associated with differentially expressed genes (DEGs). Participants in the intervention group will follow a specified dietary pattern, while the control group will maintain regular dietary habits. Peripheral blood mononuclear cells (PBMCs) will be isolated from whole blood samples via centrifugation. High-throughput RNA sequencing will analyze the transcriptome before and after dietary intervention.
Number of participants with changes in gut microbiota profile as assessed by the changes in gut microbiota diversity and composition. | 3 months
  The gut microbiota significantly impacts immune homeostasis and inflammatory skin conditions like AD. Dietary patterns influence the gut microbiome, offering a way to modulate systemic inflammation in AD. Stool samples (approx. 10mm³) will be collected from participants at baseline, day 28, day 56, and day 84 to track changes over time. Standard collection procedures will preserve microbial diversity. Participants in the intervention group will follow a specified dietary pattern, while the control group will maintain regular dietary habits. Microbial DNA will be extracted from stool samples using commercial kits, and 16S rRNA gene sequencing will identify and quantify bacterial taxa. The sequencing will assess alpha diversity (within-sample microbiota composition) and beta diversity (between-sample variation).

CONTACTS AND LOCATIONS:
Overall Officials: Fook Tim CHEW, PhD, Principal Investigator — NUS Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided